CLINICAL TRIAL: NCT03625440
Title: Acute Effects of Waterpipe Smoking on Cognitive Measures and Cardiorespiratory Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0138-16-RMB
Record Dates: First submitted 2018-05-29; First posted 2018-08-10 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Waterpipe Smoking
Keywords: cognitive tests; carboxyhemoglobin; nicotine
MeSH Terms: conditions — Water Pipe Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group - Waterpipe Smoking (Other): The Digit span test and Paced Auditory Serial Addition Test (PASAT) performed at baseline and 30minutes after waterpipe smoking.
  The Digit span test and PASAT with waterpipe smoking
  Interventions: Diagnostic Test: The Digit span test and PASAT with waterpipe smoking
- control group (Other): The Digit span test and Paced Auditory Serial Addition Test (PASAT) without waterpipe smoking, performed at 30minures apart.
  The Digit span test and PASAT without waterpipe smoking
  Interventions: Diagnostic Test: The Digit span test and PASAT without waterpipe smoking

INTERVENTIONS:
Diagnostic Test: The Digit span test and PASAT with waterpipe smoking — Cognitive tests at baseline and 30minutes after waterpipe smoking
  Arms: study group - Waterpipe Smoking
Diagnostic Test: The Digit span test and PASAT without waterpipe smoking — The Digit span test and Paced Auditory Serial Addition Test (PASAT) at baseline and 30minutes later
  Arms: control group

SUMMARY:
Title: Acute effects of waterpipe smoking (WPS) on cognitive measures and cardiorespiratory parameters

Objectives: To evaluate the acute effect of one cession of water pipe smoking on:

1. executive functions which evaluated by cognitive tests administered included the digit span subtest Wechsler Adult Intelligence Scale (WAIS)-version III hebrew battery, and the Paced Auditory Serial Addition Test (PASAT)
2. Cardiorespiratory parameters included vital signs, spirometry parameters and lung clearance index (LCI) value
3. serum carboxyhemoglobin, nicotine, and cytokines

Design: Prospective study evaluating these parameters before and after 30 minutes of water pipe smoking (WPS).

Sample size: 55 participants (35 study group, 20 control group) Participant selection: Adults subjects who regularly smoke water pipe. Intervention: Each subject will undergo evaluation including cognitive tests, Cardiorespiratory parameters, carboxy- hemoglobin levels, nicotine levels, serum cytokines levels.

All measurements will be evaluated before and after one cession of 30 minutes water pipe smoking

DETAILED DESCRIPTION:
The effect of repeated testing 30 minutes apart without water pipe smoking (WPS) was evaluated in a group of 20 volunteers (age and sex matched).

Primary outcome parameter: Change in cognitive tests scores Secondary outcome parameter:Change in Cardiorespiratory parameters included vital signs, spirometry parameters and lung clearance index (LCI) value, serum carboxyhemoglobin, nicotine, and cytokines, before and after water pipe smoking

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers aged 18 years or older who previously experienced WPS.

Exclusion Criteria:

* pregnant or lactating women
* acute viral or bacterial illness
* oral or intravenous steroid treatment in the previous two weeks
* WPS during the previous 24 hours
* cigarette smoking during the previous 6 hours
* massive exposure to fire smoke during the previous 24 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Primary outcome parameters were executive cognitive measures - The digit span test and Paced Auditory Serial Addition Test (PASAT) | Change from baseline immediately after 30 minutes of smoking
  The digit span subtest Wechsler Adult Intelligence Scale (WAIS) version III hebrew battery. Participants hear digit sequences of increasing lengths and have to recall them forward and in reversed order. Each level contains two equal number series with different numbers. Higher values represent a better outcome. Maximus score is 30 points.
  Paced Auditory Serial Addition Test (PASAT) - Single digits are presented every 3 seconds and the participant must add each new digit to the one immediately prior to it. The score is the total number correct out of 60 possible answers. Higher values represent a better outcome. Maximus score is 60 points.

SECONDARY OUTCOMES:
Heart rate | Baseline and immediately after 30 minutes of smoking
  Physiological parameter
Respiratory rate | Baseline and immediately after 30 minutes of smoking
  Physiological parameter
Blood pressure - systolic and diastolic | Baseline and immediately after 30 minutes of smoking
  Physiological parameter
Oxygen saturation | Baseline and immediately after 30 minutes of smoking
  Physiological parameter
Pulmonary parameters - Lung clearance index (LCI) | Baseline and immediately after 30 minutes of smoking
  LCI [multiple breath washouts (MBW)] measurements were performed using the Easy-One Pro, MBW Module (NDD Medical Technologies). The system consists of a side stream ultrasonic transducer for temperature- and humidity-independent sampling of the molar mass (MMss), a mainstream ultrasonic transducer for flow sampling, and a side stream infrared CO2 analyzer (DUET ETCO2 Module, Welch Allyn OEM Technologies, Beaverton OR) to correct the MMss signal for exhaled CO2. LCI was calculated as the cumulative expired volume during the washout phase divided by the functional residual capacity (FRC), which is the number of FRC turnovers required to washout the nitrogen. An increased LCI indicated more FRC turnovers required for the washout, reflecting ventilation inhomogeneity. At least three technical acceptable MBW tests were required for inclusion of the participants in the final analysis.
Pulmonary parameters - spirometry parameters | Baseline and immediately after 30 minutes of smoking
  spirometry parameters - Spirometry was performed in accordance with the American Thoracic Society/European Respiratory Society Task Force, using a KoKo spirometer (nSpire Health, Inc.; Louisville, Colorado). Each maneuver was repeated for at least three technically acceptable forced expiratory flow volume curves; the best results were used for analysis
Carboxyhemoglobin | Baseline and immediately after 30 minutes of smoking
  Carboxyhemoglobin levels were measured in venous blood samples using an Illex co-oximeter (IL-682; Instrument Laboratory; Lexington, Massachusetts)
Serum nicotine | Baseline and immediately after 30 minutes of smoking
  Serum nicotine concentrations were determined by liquid chromatography-tandem mass spectrometry, with a limit of detection (LOD) of 1ng/mL, lower limit of quantitation (LLOQ) 2ng/mL, and upper limit of quantitation (ULOQ) of 5ng/mL (Quattro micro API equipped with Waters 2795 HPLC; Waters Corp)
Serum cytokines | Baseline and immediately after 30 minutes of smoking
  The serum cytokines interleukin (IL) 2, IL-5, IL-6, IL-10, tumor necrosis factor alpha (TNFα) and transforming growth factor beta (TGF-β) were measured and analyzed using Human Inflammatory Cytokines Multi-Analyte ELISArray™ Kit [Qiagen, kit# 336161, Hilden, Germany]. The units are (pg/ml).

CONTACTS AND LOCATIONS:
Overall Officials: Lea Bentur, Prof., Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam health care campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Hakim F, Hellou E, Goldbart A, Katz R, Bentur Y, Bentur L. The acute effects of water-pipe smoking on the cardiorespiratory system. Chest. 2011 Apr;139(4):775-781. doi: 10.1378/chest.10-1833. Epub 2010 Oct 28. PMID 21030492
- [Result] Jacob P 3rd, Abu Raddaha AH, Dempsey D, Havel C, Peng M, Yu L, Benowitz NL. Nicotine, carbon monoxide, and carcinogen exposure after a single use of a water pipe. Cancer Epidemiol Biomarkers Prev. 2011 Nov;20(11):2345-53. doi: 10.1158/1055-9965.EPI-11-0545. Epub 2011 Sep 9. PMID 21908725
- [Result] Roderique JD, Josef CS, Feldman MJ, Spiess BD. A modern literature review of carbon monoxide poisoning theories, therapies, and potential targets for therapy advancement. Toxicology. 2015 Aug 6;334:45-58. doi: 10.1016/j.tox.2015.05.004. Epub 2015 May 18. PMID 25997893
- [Result] Jasper BW, Hopkins RO, Duker HV, Weaver LK. Affective outcome following carbon monoxide poisoning: a prospective longitudinal study. Cogn Behav Neurol. 2005 Jun;18(2):127-34. doi: 10.1097/01.wnn.0000160820.07836.cf. PMID 15970733
- [Result] Shihadeh A, Schubert J, Klaiany J, El Sabban M, Luch A, Saliba NA. Toxicant content, physical properties and biological activity of waterpipe tobacco smoke and its tobacco-free alternatives. Tob Control. 2015 Mar;24 Suppl 1(Suppl 1):i22-i30. doi: 10.1136/tobaccocontrol-2014-051907. Epub 2015 Feb 9. PMID 25666550
- [Result] Bentur L, Hellou E, Goldbart A, Pillar G, Monovich E, Salameh M, Scherb I, Bentur Y. Laboratory and clinical acute effects of active and passive indoor group water-pipe (narghile) smoking. Chest. 2014 Apr;145(4):803-809. doi: 10.1378/chest.13-0960. PMID 24158379